CLINICAL TRIAL: NCT01508754
Title: Efficacy of Continuous Positive Airway Pressure (CPAP) on Blood Pressure Control of Resistant Hypertension Patients With Obstructive Sleep Apnea Syndrome (OSAS).
Brief Title: Efficacy of CPAP Treatment on Blood Pressure of Resistant Hypertension Patients With Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Financiadora de Estudos e Projetos (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Gil Fernando da Costa Mendes de Salles, PhD, Full Professor, Faculty of Medicine, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FINEP-01.08.0615.00
Record Dates: First submitted 2012-01-05; First posted 2012-01-12 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Obstructive Sleep Apnea Syndrome; Resistant Hypertension
Keywords: Continuous positive airway pressure; Ambulatory blood pressures
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Active Comparator): Treatment with Continuous Positive Airway Pressure
  Interventions: Procedure: Continuous positive airway pressure treatment
- Control (No Intervention): Usual anti-hypertensive treatment without CPAP treatment

INTERVENTIONS:
Procedure: Continuous positive airway pressure treatment — Treatment with CPAP for 6 months, pressure will be titrated during a second polysomnography.
  Arms: CPAP

SUMMARY:
The aim is to evaluate the effect of treatment with Continuous Positive Airway Pressure (CPAP) device on clinic and ambulatory blood pressures (BP) of 200 resistant hypertensive patients with moderate-severe obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
Obstructive sleep apnea syndromes (OSAS) have been demonstrated to be highly prevalent in patients with resistant hypertension (defined as uncontrolled clinic BP despite being on anti-hypertensive treatment with at least 3 drugs in optimal doses and including a diuretic). Nevertheless, the effect of treating OSAS with Continuous Positive Airway Pressure (CPAP) device on clinic and ambulatory BPs in patients with resistant hypertension is largely unknown. Hence, the primary aim of this randomized clinical trial is to evaluate the effect of CPAP on BP levels in resistant hypertensive patients with moderate-severe OSAS (defined as an apnea-hypopnea index [AHI] greater than 15 on a full polysomnographic examination). Two-hundred patients will be randomly allocated either to treatment with CPAP device plus their usual anti-hypertensive treatment or to continue their usual treatment alone for 6 months. Clinic and 24-hour ambulatory BP monitoring, laboratory evaluation (including microalbuminuria and aldosterone-to-renin ratio), 24-hour Holter monitoring, ergospirometric treadmill test, and carotid-femoral pulse wave velocity measurement will be performed before and after the 6-month treatment, with the observers blinded to the allocation group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resistant hypertension and moderate-severe obstructive sleep apnea syndrome

Exclusion Criteria:

* Older than 80 years
* Pregnant women
* Non-adherent to anti-hypertensive treatment
* Severe cognitive deficits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
clinic and ambulatory blood pressures | 6 months
  Clinic and ambulatory blood pressures (during 24-hour ambulatory blood pressure monitoring, which included both daytime and nighttime blood pressures, as well as the nocturnal dipping pattern).

SECONDARY OUTCOMES:
Microalbuminuria | 6 months
  Urinary albumin excretion rate on 24-hour urine collection
Aldosterone excess measurements | 6 months
  Serum aldosterone concentration, plasma renin activity, aldosterone-to-renin ratio and 24-hour urinary aldosterone excretion.
Arterial stiffness | 6 months
  Carotid-femoral pulse wave velocity and aortic pulse wave contour analysis (which include aortic systolic and pulse pressure and augmentation index)
Autonomic system measurements | 6 months
  Measures of autonomic system balance derived from 24-hour Holter monitoring, which includes heart rate variability on time and frequency domains.
Cardiorespiratory fitness | 6 months
  Cardiorespiratory fitness by 6 min walking test with maximum oxigen consumption measurement and by complete ergospirometric treadmill test.

CONTACTS AND LOCATIONS:
Overall Officials: Gil F Salles, PhD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, federal University of Rio de Janeiro
Locations (1):
- Program of Arterial Hypertension, University Hospital Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Goodfriend TL, Calhoun DA. Resistant hypertension, obesity, sleep apnea, and aldosterone: theory and therapy. Hypertension. 2004 Mar;43(3):518-24. doi: 10.1161/01.HYP.0000116223.97436.e5. Epub 2004 Jan 19. PMID 14732721
- [Background] Logan AG, Perlikowski SM, Mente A, Tisler A, Tkacova R, Niroumand M, Leung RS, Bradley TD. High prevalence of unrecognized sleep apnoea in drug-resistant hypertension. J Hypertens. 2001 Dec;19(12):2271-7. doi: 10.1097/00004872-200112000-00022. PMID 11725173
- [Background] Lavie P, Hoffstein V. Sleep apnea syndrome: a possible contributing factor to resistant. Sleep. 2001 Sep 15;24(6):721-5. doi: 10.1093/sleep/24.6.721. PMID 11560187
- [Background] Alajmi M, Mulgrew AT, Fox J, Davidson W, Schulzer M, Mak E, Ryan CF, Fleetham J, Choi P, Ayas NT. Impact of continuous positive airway pressure therapy on blood pressure in patients with obstructive sleep apnea hypopnea: a meta-analysis of randomized controlled trials. Lung. 2007 Mar-Apr;185(2):67-72. doi: 10.1007/s00408-006-0117-x. Epub 2007 Mar 28. PMID 17393240
- [Background] Haentjens P, Van Meerhaeghe A, Moscariello A, De Weerdt S, Poppe K, Dupont A, Velkeniers B. The impact of continuous positive airway pressure on blood pressure in patients with obstructive sleep apnea syndrome: evidence from a meta-analysis of placebo-controlled randomized trials. Arch Intern Med. 2007 Apr 23;167(8):757-64. doi: 10.1001/archinte.167.8.757. PMID 17452537
- [Background] Duran-Cantolla J, Aizpuru F, Montserrat JM, Ballester E, Teran-Santos J, Aguirregomoscorta JI, Gonzalez M, Lloberes P, Masa JF, De La Pena M, Carrizo S, Mayos M, Barbe F; Spanish Sleep and Breathing Group. Continuous positive airway pressure as treatment for systemic hypertension in people with obstructive sleep apnoea: randomised controlled trial. BMJ. 2010 Nov 24;341:c5991. doi: 10.1136/bmj.c5991. PMID 21106625
- [Background] Lozano L, Tovar JL, Sampol G, Romero O, Jurado MJ, Segarra A, Espinel E, Rios J, Untoria MD, Lloberes P. Continuous positive airway pressure treatment in sleep apnea patients with resistant hypertension: a randomized, controlled trial. J Hypertens. 2010 Oct;28(10):2161-8. doi: 10.1097/HJH.0b013e32833b9c63. PMID 20577130
- [Derived] Cardoso CRL, Roderjan CN, Cavalcanti AH, Cortez AF, Muxfeldt ES, Salles GF. Effects of continuous positive airway pressure treatment on aortic stiffness in patients with resistant hypertension and obstructive sleep apnea: A randomized controlled trial. J Sleep Res. 2020 Aug;29(4):e12990. doi: 10.1111/jsr.12990. Epub 2020 Feb 12. PMID 32048379
- [Derived] de Souza F, Muxfeldt ES, Margallo V, Cortez AF, Cavalcanti AH, Salles GF. Effects of continuous positive airway pressure treatment on aldosterone excretion in patients with obstructive sleep apnoea and resistant hypertension: a randomized controlled trial. J Hypertens. 2017 Apr;35(4):837-844. doi: 10.1097/HJH.0000000000001254. PMID 28129246
- [Derived] Muxfeldt ES, Margallo V, Costa LM, Guimaraes G, Cavalcante AH, Azevedo JC, de Souza F, Cardoso CR, Salles GF. Effects of continuous positive airway pressure treatment on clinic and ambulatory blood pressures in patients with obstructive sleep apnea and resistant hypertension: a randomized controlled trial. Hypertension. 2015 Apr;65(4):736-42. doi: 10.1161/HYPERTENSIONAHA.114.04852. Epub 2015 Jan 19. PMID 25601933
- See also: Related Info — http://www.prohart.hucff.ufrj.br